CLINICAL TRIAL: NCT03316391
Title: Prospective Study : Association Between Pococyturia and Pre-eclampsia Severity
Brief Title: Association Between Pococyturia and Pre-eclampsia Severity
Acronym: PEPOD2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0517
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pre-eclampsia: Patients in hospital for pre-eclampsia at the Hopital Femme-Mère-Enfant
  Interventions: Other: Dosage of urinary podocyturia

INTERVENTIONS:
Other: Dosage of urinary podocyturia — Dosage of urinary podocyturia at admission, delivery and post-partum visit

SUMMARY:
Pre-eclampsia is an hypertensive disorder appearing during pregnancy, inducing serious maternal, fetal and neonatal mortality and morbidity. Twenty four hours proteinuria is a key element to define pre-eclampsia severity but is delaying the result by 24 hours and constraining for the patient. A simple and rapid indicator for severe preeclampsia would help clinicians to make appropriate decision in patient management. We hypothesized that urinary podocyturia is correlated to preeclampsia severity. This is a prospective, non-interventional, monocentric study.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 years or more
* single pregnancy
* admission for pre-eclampsia
* patient receiving information and non-opposition to participate

Exclusion Criteria:

* multiple pregnancy
* in utero fetal demise excepted if associated with pre-eclampsia
* antecedent of nephropathy
* fetal malformation, chromosomal anomalies
* inability to understand information provided
* prisoner or under administrative supervision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients in hospital for pre-eclampsia at the Hopital Femme-Mère-Enfant
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Severity of pre-eclampsia | at childbirth (maximum 10 months)
  Severe preeclampsia is defined by preeclampsia with at least one of the following criteria :
  * severe hypertension (PAS ≥ 160 mmHg et/ou PAD ≥ 110 mmHg)
  * Renal impairment with: oliguria <500 ml / 24h or creatinine> 135 μmol / L or proteinuria> 5 g/d
  * acute lung edema or persistent epigastric bar or HELLP syndrome
  * eclampsia or rebellious neurological disorders (visual disturbances, polykinetic ROT, headache),
  * thrombocytopenia <100 G / L
  * Retro Placental Hematoma (HRP) or fetal repercussion.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de gynécologie-obstétrique, Pierre-Bénite, Rhône
  - Department of obstetrics, Femme Mère Enfant Hospital, Lyon, France, Bron

IPD SHARING:
Plan to Share IPD: No